CLINICAL TRIAL: NCT00326443
Title: Phase I Randomized, Double-Blind, Heterologous Prime-Boost Study of the Safety and Immunogenicity of Vi Polysaccharide Typhoid Vaccine After Priming by Live Attenuated Oral Vi+ Salmonella Typhi Strain CVD 909
Brief Title: CVD 909 Vi Prime Boost Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0009; Typhoid CVD 36000
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2010-02

CONDITIONS: Typhoid Fever
Keywords: Salmonella, vaccine, typhoid fever, S. Typhi
MeSH Terms: conditions — Typhoid Fever | interventions — Polysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 14 subjects Oral CVD 909 with buffer on Day 0. Parental Vi polysaccharide vaccine on Day 21.
  Interventions: Biological: CVD 909; Biological: Vi Polysaccharide
- 2 (Placebo Comparator): 14 subjects oral buffer placebo. Parental Vi polysaccharide vaccine on Day 21.
  Interventions: Drug: Placebo; Biological: Vi Polysaccharide

INTERVENTIONS:
Biological: CVD 909 — 5 X 10^9 CFU of oral S. Typhi vaccine strain CVD 909 with buffer administered on Day 0.
  Arms: 1
Drug: Placebo — Buffer placebo administered on Day 0.
  Arms: 2
Biological: Vi Polysaccharide — 25 micrograms (0.5 ml) of licensed purified Vi polysaccharide vaccine on Day 21.

SUMMARY:
The purpose of this research study is to see if giving a typhoid vaccine by mouth (an experimental vaccine, CVD 909) before giving a vaccine shot (Typhim Vi) will result in a better immune response than giving Typhim Vi vaccine by itself. Another purpose is to see whether CVD 909 is safe. Typhim Vi has been shown to be safe and effective in preventing typhoid fever in older children and adults, but it does not work in children under age 2. Scientists at the University of Maryland think that young children could respond to Typhim Vi if they were given a dose of the other typhoid vaccine by mouth before they are given the Typhim Vi shot. Twenty-eight healthy adult volunteers, ages 18-40 years, will take part in this study. Study participation will last for up to 63 weeks, but most of the study visits will be in the first 6 weeks. Blood samples will be collected approximately 13 times. Four stool samples will be collected. Some volunteers may be followed for an additional 4 years.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, heterologous prime-boost study of the safety and immunogenicity of Vi polysaccharide typhoid vaccine after priming by live, attenuated oral Vi+ Salmonella Typhi strain CVD 909. The primary study objective is to determine the phase 1 safety of the prime-boost regimen of priming with CVD 909, a live attenuated Vi+ S. Typhi strain, followed by boosting with licensed parenteral Vi polysaccharide vaccine in healthy adult volunteers. The secondary objective is to compare the immunogenicity of licensed parenteral Vi polysaccharide vaccine in volunteers primed with a single oral dose of CVD 909 and in volunteers who are not primed with the oral vaccine. The outcome measures of interest are the seroconversion rate and titer of serum IgG anti-Vi antibodies, the timing of development and longevity of serum anti-Vi antibodies, the subclasses and avidity of antibodies developed, and the memory B and T cell responses elicited. The following immunologic outcome measures will be sought: rate and timing of seroconversion in each study arm after receiving Vi polysaccharide and analysis of immunoglobulin subclasses and avidity. This will assess the presence of priming and the rapidity of the anamnestic response. A successful priming would accelerate the response to the boost (Day 7 after Vi vaccine), and this response is expected to be more balanced, inducing both Th1/Th2-type immunity evidenced by the induction of both IgG1 and IgG2; geometric mean titer (GMT) of serum IgG anti-Vi antibodies on Days 7, 14, 21, and 35 post-Vi (Days 28, 35, 42, and 84 of the study). This will assess magnitude of response (another measure of priming); GMT of serum IgG Vi antibody in each study arm at multiple later time points up to 1 year after receiving parenteral Vi (week 55 of the study). This will assess the quality and duration of the antibodies; and peripheral blood mononuclear cells will be collected to measure cytokine production and cytotoxic T lymphocyte (CTL) activity, as well as the induction and maintenance of B and T cell memory responses and homing potential of antibody secreting cells (ASC) and T cells depending on cell numbers. Twenty-eight healthy adult volunteers, 18-40 years of age and from the Baltimore community, will be recruited to participate in this study, which will be conducted at the Center for Vaccine Development (CVD), University of Maryland School of Medicine. The volunteers will be randomized to receive either 5x10^9 colony forming units of CVD 909 with buffer or buffer placebo alone. Three weeks later, all volunteers will receive 25 micrograms (0.5 ml) of licensed purified Vi polysaccharide vaccine by the intramuscular route. Blood for serum and antibody secreting cell responses to Vi, S. Typhi LPS, and O antigen will be drawn before and after the Vi boost. The patient participation duration is up to 63 weeks, with the option for prolonged immunologic follow-up for 4 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years, inclusive.
* Good general health as determined by a screening evaluation within 30 days before administration of CVD 909 or placebo.
* Expressed interest and availability to fulfill the study requirements.
* Informed, written consent.
* Agrees not to participate in another investigational vaccine or drug trial for the first 84 days of this study.
* Agrees not to become pregnant from the time of study enrollment until at least 56 days after the administration of CVD 909 or placebo; if a woman is sexually active and capable of conception (i.e., no history of hysterectomy or tubal ligation), she must agree to use hormonal or barrier birth control. A woman is eligible if she is monogamous with a vasectomized male.

Exclusion Criteria:

* History of any of the following medical illnesses:
* Gall bladder disease or gall stones without cholecystectomy
* Diabetes
* Cancer
* Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
* Unconsciousness
* Seizures (other than febrile seizures as a child less than 5 years old)
* Recurrent infections (more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
* Any current illness requiring daily medication other than vitamins, birth control, or stable regimen of anti-histamine medication for hay fever or anti-depressant
* History of the following types of abdominal surgery:
* Any major gastrointestinal surgery (e.g., intestinal resection or splenectomy)
* A laparotomy for any reason (e.g., hysterectomy, Caesarean section, appendectomy, or herniorrhaphy) within the last 3 years
* Laparoscopic abdominal surgery within the past year
* A large abdominal scar of unclear origin
* Evidence of gastrointestinal disease, as indicated by any of the following:
* Usual bowel habit of more than 3 bowel movements each day
* Recurrent diarrhea (greater than 5 episodes during the past 6 months, each lasting at least 3 days, with at least one week between episodes)
* Lactose intolerance
* Frequent indigestion or heartburn that requires daily antacids or other medical therapy
* Diagnosed by a doctor as having irritable bowel disease, Crohn's disease, ulcerative colitis, celiac disease, stomach or intestinal ulcers in the past 10 years
* Blood in the stool during the past year (other than occasional small amount from straining)
* Any clinically significant abnormality detected on physical examination, including:
* Murmur (other than a functional murmur)
* Focal neurological deficit suggesting a pathologic process
* Hepatosplenomegaly
* Lymphadenopathy
* Jaundice
* Hypertension (BP greater than 150/90 mm Hg on two separate days) or hypotension (BP less than 85/55 mm Hg)
* Any lab abnormality, as listed below:
* WBC outside the normal range
* Hemoglobin outside the normal range
* Platelet count outside the normal range
* Creatinine outside the normal range
* Fasting glucose greater than 115 mg/dl (if screening greater than 115 mg/dl)
* AST or ALT outside the normal range (may be repeated once if outside this limit)
* Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen
* Stool culture positive for Salmonella spp, Shigella spp, Campylobacter jejuni, V. cholerae, or pathogenic protozoa
* For women, positive serum pregnancy test within 7 days and urine pregnancy test within 24 hours of administering CVD 909 and within 24 hours of administering Vi vaccine
* Nursing mother
* Oral temperature greater than 37.8ºC or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis on the day of administration of CVD 909 or placebo
* Immunization against typhoid fever or history of typhoid fever
* Allergy to quinolones (including ciprofloxacin) or sulfa drugs (Including trimethoprim/sulfamethoxazole)
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Failure to pass written examination about study purpose, background, and procedures (70% correct answers required to pass)
* Receipt of an investigational vaccine or drug within 28 days before administration of CVD 909
* Commercial food-handlers
* Health care workers who are engaged in patient care during the study
* Day care providers
* Subject with a household contact who is less than 2 years of age, who is immunocompromised or pregnant, or who works as a commercial food-handler
* Use of antibiotics within 7 days of CVD 909 or placebo vaccination
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety: determined by symptom diaries, interim medical histories obtained by interview, by blood and stool cultures, and by clinical laboratory tests. | During the 1st 14 days after ingestion of CVD 909 vaccine or placebo, during the 3 days after receiving parenteral Typhim Vi vaccine at Day 24, and interim medical history for safety at Day 42.

SECONDARY OUTCOMES:
Immunogenicity: assessed by specific antibody secreting cell assays. | Days 0 and 10 after oral administration of CVD 909 and Days 0 and 7 after administration of parenteral Vi.
The timing of development and longevity of serum anti-Vi antibodies. | Days 0 and 10 after oral administration of CVD 909 and Days 0 and 7 after administration of parenteral Vi.
The subclasses and avidity of antibodies developed. | Days 0 and 10 after oral administration of CVD 909 and Days 0 and 7 after administration of parenteral Vi.
Seroconversion rate and titer of serum IgG anti-Vi antibodies. | Days 0, 10, 14+/-2, 21+/-2, 28+/-2, 35+/-2, 42+/-2, and 84+/-7 and at 29+/-2 weeks and 55+/- 4 weeks, and every 6 months for 4 years for volunteers who remain seropositive at week 55 and agree to continue participation in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Wahid R, Zafar SJ, McArthur MA, Pasetti MF, Levine MM, Sztein MB. Live oral Salmonella enterica serovar Typhi vaccines Ty21a and CVD 909 induce opsonophagocytic functional antibodies in humans that cross-react with S. Paratyphi A and S. Paratyphi B. Clin Vaccine Immunol. 2014 Mar;21(3):427-34. doi: 10.1128/CVI.00786-13. Epub 2014 Jan 15. PMID 24429069